CLINICAL TRIAL: NCT03742479
Title: A Single Center, Prospective, Open-label, Clinical Trial Using Micro-injections of Transparent Hyaluronic Acid Gel (Restylane® Silk) for Rejuvenation of the Aging Cheek
Brief Title: Restylane Silk Microinjections to Cheeks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Principal Investigator, Isabella Guiha, Certified Clinical Research Coordinator, Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Silkcheek-2018-01
Record Dates: First submitted 2018-11-08; First posted 2018-11-15 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Wrinkle

STUDY DESIGN:
Intervention Model Description: Single Group, Open Label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hyaluronic Acid Microinjection (Experimental)
  Interventions: Device: Restylane® Silk

INTERVENTIONS:
Device: Restylane® Silk — Injectable Hyaluronic Acid (HA)

SUMMARY:
The objective of this study is to determine the efficacy and safety of Restylane® Silk microinjections when used in a grid-like injection pattern for the correction of fine lines to the cheeks.

DETAILED DESCRIPTION:
Silk for correction of mid to low cheek fine lines and wrinkles. Twenty (20) subjects will be enrolled. Each subject will receive Restylane® Silk to the entire cheeks. The defined area will be defined as the following: line extending from the upper margin of the nasal ala to the upper margin of the tragus, from the tragus to 1 cm above the mandibular angle, from 1 cm above the mandibular angle to 1 cm above the pre-jowl sulcus, and from 1 cm above the pre-jowl sulcus to the upper margin of the nasal ala. The injections will be delivered intradermally via multiple 0.02 cc microinjections distributed in a grid array pattern with 1-2 cm between each injection point (see figure 1; injections will extend 1 cm above the illustration). Following completion of injection treatment, manual massage will be applied to the full area to promote even distribution of the product. Each subject will undergo a total of three treatment sessions, one month apart, day 1, week 4, and week 8. The maximum amount of Restylane to be used per treatments session/per cheek is 1.5cc (not to exceed a total of 9 cc) per treated patient. Three-dimensional digital photography utilizing the Vectra 3D System (Canfield) will be utilized to document pre-treatment status, sites of injection, and post-treatment effect. Subjects will be followed up at 4 weeks, 8 weeks, post-treatment day 90, and day 180. Objective measures of efficacy will be me performed pre-treatment, at day 90 and 180.

ELIGIBILITY:
Inclusion Criteria:

b. Symmetrical visible sign of aging involving at least a 9 cm2 area of the mid to low cheeks.

c. Must be willing to give and sign a HIPPA form, photo consent and informed consent form.

d. Must be willing to comply with study dosing and complete the entire course of the study.

e. Female patients will be either of non-childbearing potential defined as:

1. Having no uterus 2. No menses for at least 12 months. Or; (WOCBP) women of childbearing potential must agree to use an effective method of birth control during the course of the study, such as:

1. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device
2. Intrauterine coil
3. Bilateral tubal ligation
4. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
5. Abstinence (If practicing abstinence must agree to use barrier method described above (4) if becomes sexually active).
6. Vasectomized partner (must agree to use barrier method described above (4) if becomes sexually active with un-vasectomized).

   f. Negative urine pregnancy test results Baseline prior to study entry (if applicable)

   Exclusion Criteria:
   1. Pregnant, planning pregnancy during the course of the study or breastfeeding
   2. Extremely Severe aging face with extensive photodamage
   3. Previous use of any form of soft tissue augmentation in the treatment area within the past 12 months
   4. Pre-existing medical or dermatologic condition in the treatment area that may affect the treatment or interpretation of treatment effect (at investigator discretion)
   5. Presence of tattoo and/or scar in the treatment area that in the investigators opinion would interfere with study assessments
   6. Use of oral/topical retinoids within 1 month of Baseline
   7. Previous use of botulinum toxins in the treatment area within the past 6 months
   8. Previous surgical procedure in the treatment area within the past 12 months
   9. Presence or evidence of any conditions that in the opinion of the investigator might impede the subject's ability to give consent or comply with protocol requirements.
   10. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study
   11. History of non-compliance with clinical research protocols
   12. Ablative laser resurfacing to on their face within 12 months
   13. Non-ablative laser or light procedures to their face within the past 3 months
   14. Known allergy to Restylane® Silk or any of its constituents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Investigator five point global aesthetic improvement score | Baseline to 6 - Months Post Final Treatment
  Change in Investigator five point global aesthetic improvement score from Baseline at all follow up visits through month 6 using Investogator's Global Aesthetic Improvement Scale
Cutometer Measured Skin Elaticity | Baseline to 6 - Months Post Final Treatment
  Change in elasticity from baseline to the last visit measured using a Cutometer
Hydrometer measured Transepidermal Water Loss | Baseline to 6 - Months Post Final Treatment
  Change in transepidermal waterloss from baseline to the last visit measured using a hydrometer.

SECONDARY OUTCOMES:
Safety - Injection Site Adverse Events | Baseline to 6 - Months Post Final Treatment
  At each follow up visit, any adverse effects such as but not limited to bruising, erythema, swelling, pain, tenderness, itching, dysesthesia, and nodularity will be recorded descriptively.

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No